CLINICAL TRIAL: NCT02749214
Title: Defining a Parkinson's Disease (PD) -Specific Breath Fingerprint of Underlying Inflammatory and Neurodegenerative Processes
Brief Title: Defining a PD-specific Breath Fingerprint of Underlying Inflammatory and Neurodegenerative Processes
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Malu Tansey, Associate Professor, Emory University
Other Study IDs: IRB00086732
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath samples will be collected to analyze for breath volatile organic compounds (BVOC). Peripheral blood samples will also be collected and analyzed for inflammatory proteins.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's Disease (PD): Participant's with Parkinson's Disease will provide peripheral blood and breath samples. Participants will also be asked to complete a neurologic exam and questionnaires.
  Interventions: Other: Blood Sample Collection; Other: Breath Sample Collection
- Healthy Control: Age and gender-matched healthy controls will provide peripheral blood and breath samples. Participants will also be asked to complete a neurologic exam and questionnaires.
  Interventions: Other: Blood Sample Collection; Other: Breath Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Participants will have two to three tablespoons (30 cc) of peripheral blood drawn to test for inflammatory markers.
Other: Breath Sample Collection — Participants will be asked to breathe into the Breath Sampler containing a rapid passive volatile organic compounds (VOC) sampling device. A disposable mouthpiece is placed over a portion of the sampler where the participant placed his/her mouth. The mouthpiece will be disposed of after each use and a new one will be used for each participant. Prior to sample collection, the participant will be asked to rinse his/her mouth with water. Then the participant will breathe deeply into the sampler five times with breaths being five minutes apart to collect the alveolar breath.

SUMMARY:
The purpose of this study is to determine the potential for a Parkinson's Disease (PD) -specific breath signature as a non-invasive screening tool for identifying PD patients with inflammation, tracking the progression of disease, and responsiveness to various therapeutic interventions, in particular anti-inflammatory or immunomodulatory therapies. Neurological disorders include any disorder involving the brain or the nervous system, for example memory disorders, stroke, movement disorders and many other conditions.

The study will lay the foundation for future studies in which breath fingerprinting could be used as a screening technique. Investigators will also be looking at how the breath fingerprint correlates with inflammatory proteins in the blood.

DETAILED DESCRIPTION:
The purpose of this study is to determine the potential for a Parkinson's Disease (PD) -specific breath signature as a non-invasive screening tool for identifying PD patients with inflammation, tracking the progression of disease, and responsiveness to various therapeutic interventions, in particular anti-inflammatory or immunomodulatory therapies. Neurological disorders include any disorder involving the brain or the nervous system, for example memory disorders, stroke, movement disorders and many other conditions.

The study will lay the foundation for future studies in which breath fingerprinting could be used as a screening technique. Investigators will also be looking at how the breath fingerprint correlates with inflammatory proteins in the blood.

Investigators will determine how molecules in human breath can define a "breath signature" that can be associated with neurological disorders like Parkinson's disease. The long-term goal of this study is to use blood inflammatory marker relationships and Breath Analytical Approach to identify individuals at risk for development of neurologic disorders and to monitor the effects of immune interventions on the rate of disease progression.

The study team will recruit a total of 100 participants: 50 early stage (defined by a Hohn & Yahr Stages 1-2), non-smoking Parkinson's Disease patients from among the Emory Movement Disorders Clinic and 50 age and sex-matched healthy controls (HC). Investigators will recruit six to eight participants per month over an 18-month time period.

ELIGIBILITY:
Participants with Parkinson's Disease (PD)

Inclusion Criteria:

* Must be capable of providing written informed consent
* Non-smoking
* Clinical diagnosis of PD Hohn & Yahr Stages 1 and 2

Exclusion Criteria:

* Cognitively impaired to the degree that they are not able to provide consent

Healthy Controls

Inclusion Criteria:

* Must be capable of providing written informed consent
* Age matched and a family member or healthy community control

Exclusion Criteria:

* Diagnosed with cancer and/or undergoing cancer treatment.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with a clinical diagnosis of Parkinson's Disease Hohn & Yahr Stages 1 and 2 will be recruited from the Emory Movement and Disorders Clinic. Age and sex-matched healthy controls will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale Subscale II Score | Up to 15 minutes
  The Unified Parkinson's Disease Rating Scale Subscale II is a measure of self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food. Items are rated from 0 (normal) to 4 (severe). A higher total score indicates more severe disease.
Unified Parkinson's Disease Rating Scale Subscale III Score | Up to 15 minutes
  The Unified Parkinson's Disease Rating Scale Subscale III is a clinician-scored monitored motor evaluation. Items are rated from 0 (normal) to 4 (severe). A higher total score indicates more severe disease.
Modified Hoehn and Yahr Scale Score | Up to 15 minutes
  The Modified Hoehn and Yahr Scale is used to describe how the symptoms of Parkinson's disease progress. Stages of disease range from 1 to 5 where 5 is the most severe.
Overnight Questionnaire Score | Up to 15 minutes
  The Overnight Questionnaire is completed by a person living with the participant with Parkinson's Disease. Questions refer to behaviors witnessed during sleep. Questions are answered on a scale from 1 (never) to 4 (always). A higher score indicates more symptoms of sleep disruption.
Beck's Depression Scale Score | Up to 15 minutes
  The Beck's Depression Scale is a 21 one item scale used to describe how a participant has been feeling over the past two weeks. A total score between 0-21 indicates very low anxiety. A between 22-35 indicates moderate anxiety. A score that exceeds 36 indicates high anxiety.
Montreal Cognitive Assessment (MOCA) Score | Up to 10 minutes
  The Montreal Cognitive Assessment (MOCA) is a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total possible score is 30 points; a score of 26 or above is considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Malu Tansey, PhD, Principal Investigator — Emory University; Charlene W Bayer, PhD, Principal Investigator — Hygieia, Inc
Locations (1):
- The Emory Clinic Executive Park, Atlanta, Georgia, United States